CLINICAL TRIAL: NCT06516341
Title: Spatially and Temporally Resolving Predictive Biomarkers of Postoperative Recurrence and Complications in Chronic Intestinal Inflammation
Status: Recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Collaborators: IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo (Unknown); Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other); Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Pierpaolo Sileri, Professor, IRCCS Ospedale San Raffaele
Other Study IDs: PNRR-MCNT2-2023-12377779
Record Dates: First submitted 2024-07-11; First posted 2024-07-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis; Crohn Disease
Keywords: Ulcerative Colitis; Crohn Disease; Stenosis; Post-operative recurrence; IBD; Biomarker prediction; Stricturing disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect mucosal brushes (as per clinical practice) and additional volume of blood (during blood collection as per clinical practice) and feces at the time of surgery ad hoc for the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- UC patients: Patients with histologically confirmed UC undergoing intestinal resection due to stricturing disease. These patients will be divided into two groups:
  patients with (case group) and without (control group) postoperative recurrence
  Interventions: Procedure: UC patients
- CD patients: Patients with histologically confirmed CD undergoing intestinal resection due to stricturing disease. Divided into two groups: patients with (case group) and without (control group) postoperative recurrence
  Interventions: Procedure: CD patients

INTERVENTIONS:
Procedure: CD patients — The study will involve the collection of leftover surgical material after pathologist analysis, mucosal brushes, an additional volume of blood and feces of patients at the time of surgery
  Groups: CD patients
Procedure: UC patients — The study will involve the collection of leftover surgical material after pathologist analysis, mucosal brushes, an additional volume of blood and feces of patients at the time of surgery
  Groups: UC patients

SUMMARY:
A portion of patients with Inflammatory bowel disease often require surgical intervention since they do not respond to the current therapies. Besides this risk, patients may develop post-operative disease complications, and the factors beneath are far from being understood or predicted. The investigators hypothesize that some priming factors remain in the resection margin after surgery and act as a memory of the evolution of the disease, leading to the recurrence or complications. The following proposals are made:

1. defining and validating in humanized experimental models of intestinal inflammation the spatial and temporal dynamics of the postoperative complications-priming factors
2. integrating them into a machine-learning-driven model to determine risk indices of disease recurrence in IBD patients. This risk prediction model will not change the clinical decision-making process but will only be built for research. Consequently, patients enrolled in this study will be monitored and treated as per the standard of care.

This project will reveal possible causes and build methods predictive of postoperative complications ultimately resulting in changes in clinical management in the near future.

DETAILED DESCRIPTION:
A portion of patients with Inflammatory bowel disease often require surgical intervention since they do not respond to the current therapies. Besides this risk, patients may develop post-operative disease complications, and the factors beneath are far from being understood or predicted. The investigators hypothesize that some priming factors remain in the resection margin after surgery and act as a memory of the evolution of the disease, leading to the recurrence or complications. The following proposals are made:

1. defining and validating in humanized experimental models of intestinal inflammation the spatial and temporal dynamics of the postoperative complications-priming factors
2. integrating them into a machine-learning-driven model to determine risk indices of disease recurrence in IBD patients.

This risk prediction model will not change the clinical decision-making process but will only be built for research. Consequently, patients enrolled in this study will be monitored and treated as per standard of care. This project will reveal possible causes and build methods that could help predict postoperative complications ultimately resulting in changes in clinical management.

ELIGIBILITY:
Inclusion Criteria:

* adult (age >18 years) patients with histologically confirmed CD or UC undergoing intestinal resection due to stricturing disease, regardless of their current or past medical treatment;
* given that it is an observational study, also pregnant and breastfeeding patients could be included;
* able and willing to sign the informed consent.

Exclusion Criteria:

* patients <18 years or > 70 years;
* patients with unconfirmed both UC and CD diagnoses;
* patients with superimposed dysplasia or cancer diagnosis and resections for which post- operative endoscopic assessment of recurrence is not feasible;
* patients unable or unwilling to sign the informed consent.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational multicenter study with additional procedures performed on patients with an established diagnosis of UC and CD. It consists of a prospective and a retrospective part. The prospective part involves surgical leftover and blood collected at the time of surgery ad hoc for the study, without other risks for the patients. For the retrospective analysis, paraffin-embedded specimens already stored in the pathology unit from at least two years before the project starting date (from 1st August 2022 to 31st August 2024), will be used. Moreover, we will select and include in this study adult (age ≥18 years) patients with histologically confirmed CD or UC who have undergone surgery as per standard of care and whose surgical tissue- and blood-derived cell-suspensions have been previously collected for the already approved project IBD Biobank and stored at -80° C. The retrospective analysis will include IBD biobank samples collected since 1st August 2022 up to August 2024.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To define spatial, cellular, and molecular characteristics of IBD-derived intestinal samples | 6 months from surgery
  To define the spatial transcriptome of UC and CD-derived intestinal mucosa, IBD-derived tissues will be analized by spatial transcriptomics, either at molecular or at microbiota level on formalin-fixed paraffin-embedded (FFPE) tissues stored at our pathology unit.

SECONDARY OUTCOMES:
To build the predictive model of postoperative complications based on spatially and temporally resolved IBD characteristics | 6-12 months from surgery
  Other variables to be considered are CD4+ T-cells from the processing of blood
To determine the mechanism underlying post-operative complications by exploiting in-vivo (mouse) experimental models of intestinal inflammation. | 19-24 months from surgery
  At the time of surgery, feces will be collected from patients. The microbial component from the IBD surgical specimens will be isolated and injected into humanized animal models.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No